CLINICAL TRIAL: NCT06138158
Title: Improvement of Fear-avoidance Beliefs in Patients with Chronic Non-specific Low Back Pain Treated At the Non-specific Low Back Pain Treated in the Back School
Brief Title: Improvement of Fear-avoidance Beliefs in Patients with Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Las Palmas de Gran Canaria (Other)
Responsible Party: Principal Investigator, Aníbal Báez Suárez, Clinical Professor, University of Las Palmas de Gran Canaria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPainEduca
Record Dates: First submitted 2023-11-11; First posted 2023-11-18 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-08

CONDITIONS: Non Specific Low Back Pain
Keywords: Pain; School Health Promotion; Medical Education; Exercise
MeSH Terms: conditions — Pain; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exercise and Education Group (Experimental): They will perform an exercise program oriented according to the back school, as well as educational guidelines related to pain.
  Interventions: Procedure: Exercise and Education Group

INTERVENTIONS:
Procedure: Exercise and Education Group — Physical exercise and pain education

SUMMARY:
Non-specific chronic low back pain is the main cause of public spending on health care and labor, with a prevalence of 10.2%. Its therapeutic management is difficult, with moderate levels of pain and persistent disability over time, influenced by psychosocial factors, such as "fear-avoidance" beliefs. The supervised therapeutic exercise program associated with an educational component is one of the most effective interventions to reduce pain and disability in these patients, but its efficacy seems to be less if there are erroneous beliefs, avoidance attitudes, or fear of physical activity, since it makes it difficult to follow the recommendations. The Back School would address this problem, seeking to improve pain, disability and increase quality of life.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the influence of the intervention of the Back School of the Hospital Universitario Insular de Gran Canaria in reducing the levels of "fear-avoidance" beliefs in patients with non-specific chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-specific low back pain, age 18-65 years, acceptance of voluntary participation and signature of the informed consent document.
* Acceptance of voluntary participation and signature of the informed consent document.
* Sufficient oral and written knowledge of the Spanish language
* Absence of any other educational intervention at the present time.

Exclusion Criteria:

* Presence or suspicion of red flags
* Cognitive impairment
* Spinal surgery
* Intolerance to physical activity
* Litigation pending resolution
* Pregnancy or postpartum less than 6 months
* Withdrawal from the study (signature of the informed consent revocation document).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in the level of fear-avoidance beliefs. | Baseline and up to ten weeks
  This variable will be recorded using the Spanish version of the Fear-Avoidance Belief Questionnaire (FABQ).
  The FABQ contains 16 items. Each item is answered on a 7-point Likert scale (0 = strongly disagree; 6 = strongly agree). The FABQ-total represents the sum of all items (96 possible points). A higher score indicates more deeply held fear avoidance beliefs. There are two subscales within the FABQ: a subscale of Fear-Avoidance to physical activity, with 5 items (FABQ: items scoring 2, 3, 4 and 5; maximum score, 24), and another of Fear-Avoidance to work, with 11 items (FABQ: items scoring 6, 7, 9, 10, 11, 12 and 15; maximum score, 42). Its Spanish version has shown as good or better properties in the FABQ-total questionnaire than in its subscales to determine Fear-avoidance.
Change in Pain assessed by VAS | Baseline and up to ten weeks
  The instrument will be used to measure the change of pain before and after the intervention will be the Visual Analogue Scale (VAS).
  Participants will be asked to mark the level of their pain on a 100 mm, no hatched VAS scale marked at one end as "no pain" and at the other as "worst pain imaginable".

SECONDARY OUTCOMES:
Change in the level of disability | Baseline and up to ten weeks
  The Oswestry Disability Index (ODI: 0-100, higher score indicates greater disability) (28) or Oswestry Disability Questionnaire for back pain, which is a widely used and validated instrument to measure disability related to low back pain (29,30), will be used as a measuring instrument. The questionnaire is focused on physical activities and does not evaluate the psychological or affective component of low back pain.
Change in Sleep quality | Baseline and up to ten weeks
  The Pittsburgh Sleep Quality Index (PSQI) will be used. It consists of 19 self-administered questions and 5 questions assessed by the patient's partner or roommate (if available). Only the self-administered questions are included in the score.
  The higher the total score, the worse the sleep quality. Thus, a total score less than or equal to five on the Pittsburgh scale indicates that, in general, your sleep quality is optimal, while a total score greater than five suggests that you have sleep problems, of greater or lesser severity.

CONTACTS AND LOCATIONS:
Overall Officials: Sven Mikael Appelvik González, MSc, Principal Investigator — University of Las Palmas de Gran Canaria
Locations (1):
- Sven Mikael Appelvik González, Las Palmas de Gran Canaria, Las Palmas, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Delitto A, George SZ, Van Dillen L, Whitman JM, Sowa G, Shekelle P, Denninger TR, Godges JJ; Orthopaedic Section of the American Physical Therapy Association. Low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):A1-57. doi: 10.2519/jospt.2012.42.4.A1. Epub 2012 Mar 30. PMID 22466247
- [Background] National Collaborating Centre for Primary Care (UK). Low Back Pain: Early Management of Persistent Non-specific Low Back Pain [Internet]. London: Royal College of General Practitioners (UK); 2009 May. Available from http://www.ncbi.nlm.nih.gov/books/NBK11702/ PMID 20704057
- [Background] Sorensen PH, Bendix T, Manniche C, Korsholm L, Lemvigh D, Indahl A. An educational approach based on a non-injury model compared with individual symptom-based physical training in chronic LBP. A pragmatic, randomised trial with a one-year follow-up. BMC Musculoskelet Disord. 2010 Sep 17;11:212. doi: 10.1186/1471-2474-11-212. PMID 20849601